CLINICAL TRIAL: NCT03902522
Title: A Multi-center, Two-Part, Single-Arm, Open Label, 25-Week Trial With PRO 140 in Treatment-Experienced HIV-1 Subjects
Brief Title: PRO 140 in Treatment-Experienced HIV-1 Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 140_CD02_OpenLabel
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leronlimab (PRO 140) (Experimental): Subjects will be on existing ART for one week followed by PRO 140 700 mg weekly subcutaneous (SC) Inj. + existing ART for the next week. Subsequently, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  Interventions: Drug: PRO 140

INTERVENTIONS:
Drug: PRO 140 — 2 injections of PRO 140 (2 X 2 mL/inj.) Subjects who were previously enrolled and receiving 350 mg dose had the option to move to the 700mg dose for the remainder of the trial.
  Other Names: Leronlimab

SUMMARY:
The primary objectives of the trial are to assess the efficacy, clinical safety and tolerability parameters of PRO 140 in combination with failing ART (antiretroviral therapy) during the initial one-week treatment period, and in combination with Optimized Background Therapy during the subsequent 24-week treatment period.

DETAILED DESCRIPTION:
PRO 140, in combination with other antiretroviral agents, is indicated for treatment experienced adult HIV-1 patients infected with CCR5-tropic virus (virus that uses the chemokine receptor type 5 to enter the cell). These patients must demonstrate evidence of HIV-1 replication despite ongoing antiretroviral therapy and have documented genotypic or phenotypic resistance to at least one ART drug within three drug classes (or within two or more drug classes with limited treatment option). The options may be limited as a result of drug antiviral class cross-resistance, documented treatment intolerance, documented objective assessments such as renal or hepatic insufficiency (e.g. high creatinine at baseline, limiting treatment options due to potential for toxicity), past adverse reactions such as hypersensitivity reactions or neuropsychiatric issues that could limit use of currently approved drugs. Study population includes treatment-experienced HIV-infected patients with CCR5-tropic virus who demonstrates evidence of HIV-1 replication despite ongoing antiretroviral therapy with documented genotypic or phenotypic resistance to ART drugs within three drug classes (or within two drug classes with limited treatment option). The primary objectives of the trial are to assess the efficacy, clinical safety and tolerability parameters of PRO 140 in combination with failing ART during the initial one-week treatment period, and in combination with Optimized Background Therapy during the subsequent 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥18 years
2. Exclusive CCR5-tropic virus at Screening Visit as determined by Monogram Biosciences Trofile® Assay
3. Have a history of at least 3 months on current antiretroviral regimen
4. Treatment-experienced HIV-infected patients with documented genotypic or phenotypic resistance to at least one ART drug within three drug classes OR Treatment-experienced HIV-infected patients with documented genotypic or phenotypic resistance to at least one ART drug within two drug classes and have limited treatment option. The options may be limited as a result of drug antiviral class cross-resistance, documented treatment intolerance, documented objective assessments such as renal or hepatic insufficiency (e.g. high creatinine at baseline, limiting treatment options due to potential for toxicity), past adverse reactions such as hypersensitivity reactions or neuropsychiatric issues that could limit use of currently approved drugs.
5. Be willing to remain on treatment without any changes or additions to the OBT regimen, except for toxicity management or upon meeting criteria for treatment failure
6. Plasma HIV-1 RNA ≥ 400 copies/mL at Screening Visit as determined by Human Immunodeficiency Virus 1 (HIV-1) Quantitative, RNA (Roche Taqman® Real-Time PCR) and documented detectable viral load (HIV-1 RNA >50 copies/ml) within the last 3 months prior to Screening Visit
7. Laboratory values at Screening of:

   1. Absolute neutrophil count (ANC) ≥750/mm3
   2. Hemoglobin (Hb) ≥10.5 gm/dL (male) or ≥ 9.5 gm/dL (female)
   3. Platelets ≥75,000 /mm3
   4. Serum alanine transaminase (SGPT/ALT) <5 x upper limit of normal (ULN)
   5. Serum aspartate transaminase (SGOT/AST) <5 x ULN
   6. Bilirubin (total) <2.5 x ULN unless Gilbert's disease is present or subject is receiving atazanavir in the absence of other evidence of significant liver disease
   7. Creatinine ≤1.5 x ULN
8. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator
9. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug
10. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent Note: Subjects diagnosed with either substance dependence or substance abuse or any history of a concomitant condition (e.g., medical, psychologic, or psychiatric) may be enrolled if in the opinion of site investigator these circumstances would not interfere with the subject's successful completion of the study requirements

Exclusion Criteria:

1. Documented CXCR4-tropic virus or Dual/Mixed tropic (R5X4) virus as determined by HIV-1 tropism assay
2. Patients with no viable treatment options ( i.e., no fully active antiretroviral drug available which can be effectively combined to form a viable new OBT)
3. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma) Note: Subjects infected by the hepatitis B virus or hepatitis C virus will be eligible for the study if they have no signs of hepatic decompensation and meet the liver function tests eligibility criteria
4. Laboratory test values of ≥ grade 3 DAIDS (Division of Acquired Immune Deficiency Syndrome) laboratory abnormality with the exception of the absolute CD4+ count criterion of <200/mm3
5. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study
6. Unexplained fever or clinically significant illness within 1 week prior to the first study dose
7. Any vaccination within 2 weeks prior to the first study dose
8. Subjects weighing < 35kg
9. History of anaphylaxis to oral or parenteral drugs
10. History of Bleeding Disorder or patients on anti-coagulant therapy
11. Participation in an experimental drug trial(s) within 30 days of the Screening Visit
12. Any known allergy or antibodies to the study drug or excipients
13. Treatment with any of the following:

    1. Radiation or cytotoxic chemotherapy with 30 days prior to the screening visit
    2. Immunosuppressants within 60 days prior to the screening visit
    3. Immunomodulating agents (e.g., interleukins, interferons), hydroxyurea, or foscarnet within 60 days prior to the screening visit
    4. Oral or parenteral corticosteroids within 30 days prior to the Screening Visit. Subjects on chronic steroid therapy >5 mg/day will be excluded with the following exception:

       * Subjects on inhaled, nasal, or topical steroids will not be excluded
14. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelly, MD, Study Chair — CytoDyn, Inc.
Locations (14):
- United States (14):
  - CD02_OpenLabel Investigational Site, Palm Springs, California
  - CD02_OpenLabel Investigational Site, San Francisco, California
  - CD02_OpenLabel Investigational Site, New Haven, Connecticut
  - CD02_OpenLabel Investigational Site, Ft. Pierce, Florida
  - CD02_OpenLabel Investigational Site, Miami, Florida
  - CD02_OpenLabel Investigational Site, Orlando, Florida
  - CD02_OpenLabel Investigational Site, West Palm Beach, Florida
  - CD02_OpenLabel Investigational Site, Decatur, Georgia
  - CD02_OpenLabel Investigational Site, Chicago, Illinois
  - CD02_OpenLabel Investigational Site, Wichita, Kansas
  - CD02_OpenLabel Investigational Site, Syracuse, New York
  - CD02_OpenLabel Investigational Site, Bellaire, Texas
  - CD02_OpenLabel Investigational Site, Houston, Texas
  - CD02_OpenLabel Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Leronlimab (PRO 140): Subjects will be on existing ART (antiretrovial therapy) for one week followed by PRO 140 700 mg weekly SC Inj. + existing ART for the next week. Subsequently, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  PRO 140: 2 injections of PRO 140 (2 X 2 mL/inj.)
Period: Overall Study
Arm/Group | Leronlimab (PRO 140)
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population is defined as the set of subjects who are enrolled and have received at least one dose of PRO 140. Subjects who discontinue from the study prior to their first post-baseline assessment will be included in the ITT population and analyzed as non-responders in the primary safety analysis
Groups:
- Leronlimab (PRO 140): Subjects will be on existing ART for one week followed by PRO 140 700 mg weekly SC Inj. + existing ART for the next week. Subsequently, all subjects will enter the 24-week single-arm, open-label treatment period. During this period, all subjects will receive PRO 140 SC injection and Optimized Background Therapy.
  PRO 140: 2 injections of PRO 140 (2 X 2 mL/inj.)
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 52.7 [36 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Years since original HIV Diagnosis [Mean (Full Range); unit: Years] | 27 [10 to 46]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With ≥ 0.5 log10 Reduction in HIV-1 RNA Viral Load From Baseline at the End of the Initial 1-week Treatment Period
Description: The primary endpoint for this study is the proportion of participants with a ≥ 0.5 log10 reduction in HIV-1 RNA viral load from baseline to the end of the initial 1-week treatment period.
Time Frame: 1-week from baseline to the end of the initial PRO 140 and ART treatment period
Population: as for baseline characteristics
Measure: Number; unit: proportion of participants
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
proportion of participants | 0.80

2. Secondary Outcome: Proportion of Participants With ≥ 1 log10 Reduction in HIV-1 RNA Viral Load From Baseline at the End of the Initial 1-week Treatment Period
Description: The secondary endpoint is the proportion of participants with ≥ 1 log10 reduction in HIV-1 RNA viral load from baseline at the end of the initial 1-week treatment period
Time Frame: 1-week from baseline to the end of the initial PRO 140 and ART treatment period
Population: The Intent-to-Treat (ITT) population is defined as the set of subjects who are enrolled and have received at least one dose of PRO 140
Measure: Number; unit: proportion of participants
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
proportion of participants | 0.40

3. Secondary Outcome: Mean Change From Baseline in HIV-1 RNA Levels (log10 Copies/mL) at the End of the Initial 1-week Treatment Period
Description: The secondary endpoint is the mean change between baseline and the end of the 1-week of treatment period in HIV-1 RNA levels (log10 copies/mL) (baseline was T1, mean change was calculated between time points T1 and T2).
  If the mean change is a negative value, this indicates a reduction in viral load.
Time Frame: 1-week from baseline to the end of the initial PRO 140 and ART treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 copies per mL
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
log10 copies per mL | -0.69 (0.61)

4. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA < 400 Copies/mL at Week 25
Description: The secondary endpoint is the percentage of participants achieving HIV-1 RNA < 400 copies/mL at week 25
Time Frame: 25 weeks post-initiation of PRO 140 and existing ART treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA < 50 Copies/mL at Week 25
Description: The secondary outcome measure is the percentage of participants achieving HIV-1 RNA < 50 copies/mL at week 25
Time Frame: 25 weeks post-initiation of PRO 140 and existing ART treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
Participants | 3

6. Secondary Outcome: Mean Change From Baseline in HIV-1 RNA Levels (log10 Copies/mL)
Description: The secondary outcome measure is the mean change in HIV-1 RNA levels (log10 copies/mL) between Baseline (T1) and week 25 (T25). Baseline was T1, mean change was calculated between time points T1 and T25.
  If the mean change is a negative value, this indicates a reduction in viral load.
Time Frame: 25 weeks post-initiation of PRO 140 and existing ART treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
log10 copies/mL | -2.29 (0.63)

7. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at the End of the Initial 1-week Treatment Period
Description: The secondary outcome measure is the mean change in CD4 cell count between Baseline and the end of the initial 1-week treatment period (T2). Baseline was T1, mean change was calculated between time points T1 and T2.
Time Frame: 1-week post-initiation of PRO 140 and ART treatment.
Population: as for outcome 2
Measure: Mean (Full Range); unit: cells/uL
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
cells/uL | 37.4 [-13 to 92]

8. Secondary Outcome: Mean Change From Baseline in CD4 Cell Count at Week 23
Description: The secondary outcome measure is the mean change in CD4 cell count between Baseline (T1) and week 23 (T23)
Time Frame: 23 weeks post-initiation of PRO 140 and existing ART treatment
Population: The outcome measure stated change from baseline at week 25 but CD4 cell count data was not collected at week 25. The last week CD4 cell count was collected was week 23. Change from baseline was calculated at week 23.
Measure: Mean (Full Range); unit: cells/uL
Arm/Group | Leronlimab (PRO 140)
Number analyzed (Participants) | 5
cells/uL | 123 [3 to 254]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were assessed from T1 visit up to T25 visit (up to 32 weeks).
Description: AEs will be elicited through direct questioning and subject reports. Any abnormalities in visit evaluations, physical examination findings or laboratory results that the Investigator believes are clinically significant to the research subject and that occurred after initiation of the first study treatment (T1) will be reported as AEs.
Groups:
- Leronlimab (PRO 140) + Existing ART: Subjects received existing Anti-Retroviral Therapy (ART) and PRO 140 700 mg SC Injection (T1 - 1 week treatment period).
- Leronlimab (PRO 140) + OBT: Subjects received PRO 140 weekly SC injection and Optimized Background Therapy (OBT) (T2 - T25 - 24-week treatment period).
Arm/Group | Leronlimab (PRO 140) + Existing ART | Leronlimab (PRO 140) + OBT
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leronlimab (PRO 140) + Existing ART (N=6) | Leronlimab (PRO 140) + OBT (N=6)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leronlimab (PRO 140) + Existing ART (N=6) | Leronlimab (PRO 140) + OBT (N=6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
According to the information provided by contract research organization (CRO), lab data for CD4 cell count was not collected at week 25. This outcome measure could not be reported in a data table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03902522/Prot_001.pdf